CLINICAL TRIAL: NCT00682604
Title: Community Health Agents From East Zone of Sao Paulo City, Brazil: A Look at Their Nutritional Status and Food Intake
Brief Title: The Nutritional Status and Food Intake of Community Health Agents
Status: Completed | Type: Observational
Sponsor: Unidade Itaquera (Other)
Responsible Party: Alexandra Corrêa de Freitas, UItaquera
Other Study IDs: UItaquera
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Nutritional and Metabolic Diseases
Keywords: Family Health Program; Food consumption; Nutritional status
MeSH Terms: conditions — Nutritional and Metabolic Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This research had as a goal to characterize the social demographic profile, nutritional status, the presence of chronic non-transmissible diseases and food intake of the community health agents who belong to five family health units in the east zone of Sao Paulo City.

DETAILED DESCRIPTION:
It's a descriptive, exploratory and quantitative study developed among 88 individual.

ELIGIBILITY:
Inclusion Criteria:

* Be an agent comunnity health who belong in the family health unit choosed to participate of this study;
* Assign the autorization to participate of the study;
* Answer a questionary of health, social demographic profile and food intake.

Exclusion Criteria:

* Refuse to participate or assign the autorization;
* Don´t answer the questionary of health and food intake;
* Don´t participate of the nutricional status evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community health agents from East Zone of Sao Paulo City, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2006-09; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra C. Freitas, Principal Investigator — Faculdade Santa Marcelina - Unidade Itaquera
Locations (1):
- Faculdade Santsa Marcelina - Unidade Itaquera, São Paulo, São Paulo, Brazil